CLINICAL TRIAL: NCT03265808
Title: A Phase I/II, Prospective, Randomized, Double-Blind, PlAcebo-ControLled Trial to EvAluate the Efficacy of Allogeneic HUman Mesenchymal Stem Cell InfusioN Versus Placebo in Subjects With Alcohol Use Disorder and Major DepreSsion.(ALAUNUS)
Brief Title: Allogeneic Human Mesenchymal Stem Cell Infusion vs Placebo in Alcohol Use Disorder and Major Depression.
Acronym: Alaunus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ihsan M Salloum, MD, MPH (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Ihsan M Salloum, MD, MPH, Professor, University of Texas Rio Grande Valley
Organization: University of Texas Rio Grande Valley (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170674; 1R01AA024933-01A1 (NIH)
Record Dates: First submitted 2017-08-16; First posted 2017-08-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; Alcohol Use Disorder
Keywords: stem cells
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- allogeneic human mesenchymal stem cells (allo-hMSCs) (Experimental): Participants will be treated with a single administration of allogeneic hMSCs: 100 x 10^6 (100 million) allo-hMSCs of cells delivered via a single peripheral intravenous infusion.
  Interventions: Drug: allogeneic human mesenchymal stem cells (allo-hMSCs)
- Placebo (Placebo Comparator): Participants will be treated with a placebo administration consisting of 1% human albumin serum in Plasma-Lyte A delivered via a single peripheral intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: allogeneic human mesenchymal stem cells (allo-hMSCs) — Single administration of allogeneic hMSCs: 100 x 106 (100 million) allo-hMSCs of cells delivered via a single peripheral intravenous infusion.
  Arms: allogeneic human mesenchymal stem cells (allo-hMSCs)
Drug: Placebo — Placebo administration consisting of 1% human albumin serum in Plasma-Lyte A delivered via a single peripheral intravenous infusion.
  Arms: Placebo

SUMMARY:
The purpose of this study is to look at the safety of a study treatment with stem cells in Alcohol Use Disorder And Major Depression (AUD-MD) subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind placebo-controlled study of allogeneic human mesenchymal stem cell in subjects with comorbid Alcohol Use Disorder And Major Depression (AUD-MD). 80 subjects will be randomized (1:1) to active treatment vs. placebo an followed weekly for 12 weeks and then every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Subjects age >18 and <75 years at the time of signing the Informed Consent Form.
3. Diagnostic and Statistical Manual of Mental Disorder-5 criteria for Alcohol Urge Questionnaire (moderate or severe defined as meeting 4 or more of the 11 criteria) AND a concurrent Diagnostic and Statistical Manual of Mental Disorder-5 recurrent unipolar major depression with HRSD-25 score of 18 or above.
4. A history of a depressive episode occurring or persisting during a period of one-month abstinence.
5. Participants should express the desire to reduce or stop alcohol consumption, report 28 or more standard drinks (SD) per week for males or 21 for females over four weeks during the 90 days preceding study enrollment.
6. Increased inflammation ([serum C-reactive protein] ≥3.0 mg/L.
7. Agree to taper and discontinue antidepressant medications during the 12-week trial.
8. Able to provide informed consent and comply with study procedures.
9. Able to read English and understand study instruments.
10. Entry criteria for depression and alcohol use disorder (moderate or severe) will be established using the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (SCID) for categorical diagnosis.
11. Have a score of ≥18 on the Hamilton Depression Rating Scale for Depression (HAM-D).

Exclusion Criteria:

1. Acute suicidality.
2. Any lifetime history of bipolar disorder, schizophrenia, or schizoaffective disorder.
3. Active psychotic disorder, eating disorder, or substance use disorder except for alcohol and tobacco or "mild" cannabis use disorder within 6 months of enrollment.
4. Any lifetime history of autoimmune or immunodeficiency syndrome.
5. Treatment with any psychotropic (including hypnotic), steroidal, or anti-inflammatory medication (including NSAIDs) within 2 weeks of treatment randomization (6 weeks for fluoxetine).
6. Any current use of medication that affect alcohol consumption such as acamprosate, disulfiram, naltrexone (po or IM), topiramate, or sedative-hypnotics including benzodiazepines or any psychostimulant.
7. Being enrolled in an alcohol treatment program (self-help groups participation such as Alcoholics Anonymous or Dual Diagnosis self-help are allowed).
8. Active medical condition that could cause or exacerbate depressive symptoms (e.g., hypothyroidism, anemia).
9. Currently pregnant or breast-feeding.
10. Lack of use of a reliable means of contraception methods. (Female subjects of childbearing potential must undergo a serum or urine pregnancy test at screening and within 36 hours prior to infusion.)
11. First major depressive episode after 50 years of age.
12. Any evidence of current infection including serum positive for HIV, hepatitis BsAg or Viremic hepatitis.
13. Medical conditions with known autoimmune or inflammatory mechanisms including any chronic allergic condition.
14. Positive urine screens for any drug of abuse other than cannabis at baseline.
15. Inability to read or understand study forms or informed consent or the presence of any other conditions or factors, which in the opinion of the investigator would make the patient unsuitable for study participation.
16. Prior history of a suicide attempt, within the past year.
17. Have hypersensitivity to dimethyl sulfoxide (DMSO).
18. Have a clinical history of malignancy within 3 years (i.e., subjects with prior malignancy must be disease free for 3 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma.
19. Be serum positive for HIV, hepatitis BsAg or Viremic hepatitis C.
20. Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Incident of treatment emergent-serious adverse events | One month post-infusion
  Incidence of any treatment-emergent serious adverse events, defined as a composite of acute suicidality and hospitalization for suicide attempts.

SECONDARY OUTCOMES:
Change in serum concentrations of high sensitivity C-reactive protein. | Baseline, 12 weeks
  Change in serum concentrations of high sensitivity C-reactive protein. A serum sample will be collected to assess the change.
Change in serum concentrations of inflammatory biomarkers | Baseline, 12 weeks
  Change in serum concentrations of inflammatory biomarkers, such as in TNF alpha and interleukin-6. A serum sample will be collected to assess the change.
Change in depressive symptoms as assessed by MADRS | Baseline, 12 weeks
  Montgomery and Asberg Depression Rating Scale (MADRS) is a ten item questionnaire with a total score ranging from 0-60 with a higher score indicating higher depressive symptoms.
Change in Depressive symptoms as assessed by CGI | Baseline, 12 weeks
  Clinical Global Improvement (CGI) is rated on a 7 point scale ranging from 1 (very much improved) to 7 (very much worse).
Change in quantity of alcohol use as assessed by TLFB | Baseline, 12 weeks
  30-day self report Timeline Follow Back (TLFB) questionnaire will be used to assess daily alcohol use.
Change in frequency of alcohol use as assessed by TLFB | Baseline, 12 weeks
  30-day self report Timeline Follow Back (TLFB) questionnaire will be used to assess frequency of daily alcohol use.
Change in Anhedonia as measured by SHAPS | Baseline, 12 weeks
  Snaith Hamilton Pleasure Scale (SHAPS) is a 14 item questionnaire with a total score ranging from 0-56 with a higher score indicating increased anhedonic symptoms.
Change in cravings as assessed by AUQ | Baseline, 12 weeks
  Alcohol Urge Questionnaire (AUQ) is an 8 item questionnaire with total score ranging from 8-56 with a high score indicating increased cravings .
Change in cravings as assessed by OCDS | Baseline, 12 weeks
  Obsessive-Compulsive Drinking Scale (OCDS) is a 14 item questionnaire ranging from 0-56 with a higher score indicating increase cravings.
Change in cognition as assessed by BAC-A | Baseline, 12 weeks
  Brief Assessment of Cognition for Affective Disorders (BAC-A) includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed. Z-scores are calculated from composite scores. Higher z-scores are indicative of better cognitive performance, lower z-scores are indicative of lower cognitive performance. Range of z-scores anticipated to be between -3 and 3.
Change in functioning as assessed by UPSA-B | Baseline, 12 weeks
  University of California of San Diego (UCSD) Performance Based Skills Assessment (UPSA-B) questionnaire has a total score from 0-100 with a higher score indication better functioning.
Change in functioning as assessed by GAF | Baseline, 12 weeks
  Global Assessment of Functioning (GAF) questionnaire has a total score ranging from 1-100 with a higher score indicating of daily activities.
Change in quality of life as assessed by QOLI | Baseline, 12 weeks
  Quality of Life Index (QOLI) questionnaire has a total score ranging from 10-100 with a higher score indicating higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ihsan Salloum, MD, Principal Investigator — University of Texas Rio Grande Valley School of Medicine
Locations (1):
- University of Texas Rio Grande Valley School of Medicine, Harlingen, Texas, United States

IPD SHARING:
Plan to Share IPD: No